CLINICAL TRIAL: NCT06596863
Title: Association of Serum Uromodulin and DKD a Systematic Review and Meta Analysis
Brief Title: Serum Uromodulin and DN Systematic Review and Meta Analysis
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shaimaa Ibrahim Barr, Dr of Biochemistry, Tanta University
Other Study IDs: DKD serum uromodulin
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Nephropathies
Keywords: DKD, urimodulin
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Glomerular Filtration Rate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Included 862 healthy subjects as control group
  Interventions: Diagnostic Test: The association of serum uromodulin with DN; Diagnostic Test: The DN patients were divided according to the level of albumin to creatinine ratio (ACR), glomerular filtration rate (GFR), or albumin excretion rate (AER) in patients with DN
- DKD group: Included 912 patients with DN
  Interventions: Diagnostic Test: The association of serum uromodulin with DN; Diagnostic Test: The DN patients were divided according to the level of albumin to creatinine ratio (ACR), glomerular filtration rate (GFR), or albumin excretion rate (AER) in patients with DN

INTERVENTIONS:
Diagnostic Test: The association of serum uromodulin with DN — Meta analysis of association of serum uromodulin with DKD
Diagnostic Test: The DN patients were divided according to the level of albumin to creatinine ratio (ACR), glomerular filtration rate (GFR), or albumin excretion rate (AER) in patients with DN — DN patients were divided according to the level of albumin to creatinine ratio (ACR), glomerular filtration rate (GFR), or albumin excretion rate (AER) in patients with DN

SUMMARY:
Several studies have investigated the association between the changes of serum uromodulin and diabetic nephropathy (DN). However, the results are still controversial. Hence, this meta-analysis aimed to evaluate the association of uromodulin with DN.

ELIGIBILITY:
Inclusion Criteria:

* Studies were included if they met the following criteria:

  1. serum level of uromodulin was determined;
  2. the samples were enrolled from diabetic patients;
  3. mean ± SD was reported for uromodulin between patients with and without DN;
  4. the level of albumin to creatinine ratio (ACR), glomerular filtration rate (GFR), or albumin excretion rate (AER) in patients with DN was determined

Exclusion Criteria:

* Studies were excluded according to the following criteria:

  1. duplicate studies;
  2. review articles;
  3. non original research articles;
  4. studies with insufficient data to extract;
  5. non-human research;
  6. studies that determined urine level of uromodulin.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The systematic search strategy retrieved 275 publications by the 4 databases (PubMed 76, Cochrane Library 11, Web of Science 107, and Scopus 81). 144 studies remained after exclusion the duplicates. After screening title and abstract 135 studies were excluded. 9 studies remained for full text and data reviewing. 4 studies of them were excluded as they didn't meet the eligibility criteria. In addition, 1 study was retrieved by manual search from Google Scholar. Finally, 6 articles were included [20-25]. The selected studies included 1774 participant
Sampling Method: Non-Probability Sample
Enrollment: 1774 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Association of serum uromodulin with DKD: asystematic review and meta analysis | may, 2024
  Evaluate the meta analysis of association of serum uromodulin in the 3 diabetic group comparing with each other and compare them to the control group and correlate these results with other kidney biomarker

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Yniversity, Tanta, Yes, Egypt

IPD SHARING:
Plan to Share IPD: No